CLINICAL TRIAL: NCT00061113
Title: Substance Dependent Teens - Impact of Treating Depression Study 1
Brief Title: Substance Dependent Teens - Impact of Treating Depression Study 1 - 1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Paula Riggs, M.D., University of Colorado Denver
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-13176-1; R01-13176-1
Record Dates: First submitted 2003-05-21; First posted 2003-05-22 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-09

CONDITIONS: Alcohol-Related Disorders; Marijuana Abuse; Substance-Related Disorders
Keywords: alcohol dependence; marijuana dependence
MeSH Terms: conditions — Alcohol-Related Disorders; Marijuana Abuse; Substance-Related Disorders; Alcoholism | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): fluoxetine + CBT
  Interventions: Drug: Fluoxetine + outpatient cognitive behavioral therapy; Drug: fluoxetine
- 2 (Placebo Comparator): placebo + CBT
  Interventions: Drug: placebo + CBT

INTERVENTIONS:
Drug: Fluoxetine + outpatient cognitive behavioral therapy — single fixed morning dose 20 mg X 15 weeks
  Other Names: Prozac
  Arms: 1
Drug: fluoxetine — 20mg, QD x 16 weeks
  Other Names: prozac
  Arms: 1
Drug: placebo + CBT — single fixed morning dose X 16 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the impact of treating depression on substance dependent teens.

DETAILED DESCRIPTION:
The primary study aim is to determine whether fluoxetine + CBT is a more effective treatment than placebo + CBT for substance outcomes, depression, and behavior problems. The current community standard of care often withholds pharmacotherapy for depression in substance abusing adolescents, since it is often assumed that their depressions may remit with SUD treatment alone. However, this is an untested hypothesis in adolescents and one that we propose to test in the current study.

ELIGIBILITY:
Inclusion Criteria:

* Must have DSM IV non bipolar Major Depressive disorder (by clinical interview), DSM IV Conduct Disorder, and Non-Tobacco Substance Disorder.

Exclusion Criteria:

* History of or current psychosis, history of psychotic depression, bipolar disorder I or II, family history of first degree relative with bipolar I, lifetime history of non-substance induced Mania/Hypomania
* Unstable chronic or serious medical illness
* Currently pregnant
* Take psychotrophic medication, past 2 months: medication or treatment for depression, clinically significant laboratory abnormality

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 126 (Actual)
Dates: Start 2001-02; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To determine whether fluoxetine + CBT is a more effective treatment than placebo + CBT for substance outcomes, depression, and behavior problems. | 16 weeks

SECONDARY OUTCOMES:
To determine if the treatment of depression with fluoxetine + CBT, in depressed adolescents with SUD and CD will be more effective than placebo + CBT in reducing substance use and improving conduct symptoms. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paula Riggs, M.D., Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Denver, Aurora, Colorado
  - 1611 South Federal Blvd., Denver, Colorado

REFERENCES:
- [Background] Deas D, Riggs P, Langenbucher J, Goldman M, Brown S. Adolescents are not adults: developmental considerations in alcohol users. Alcohol Clin Exp Res. 2000 Feb;24(2):232-7. PMID 10698377
- [Background] Davies RD, Gabbert SL, Riggs PD. Anxiety Disorders in Neurologic Illness. Curr Treat Options Neurol. 2001 Jul;3(4):333-346. doi: 10.1007/s11940-001-0038-1. PMID 11389804
- [Background] Riggs PD, Davies RD. A clinical approach to integrating treatment for adolescent depression and substance abuse. J Am Acad Child Adolesc Psychiatry. 2002 Oct;41(10):1253-5. doi: 10.1097/00004583-200210000-00016. No abstract available. PMID 12364848
- [Background] Riggs PD. Treating adolescents for substance abuse and comorbid psychiatric disorders. Sci Pract Perspect. 2003 Aug;2(1):18-29. doi: 10.1151/spp032118. PMID 18552718
- [Background] Laudenslager, M.L., Neu, M., Riggs, P., Goldstein, M., & Lohman, M. Refinements in a novel technique for collecting saliva for steroid hormone determinations. Brain Behavior, and Immunity, 17 (3), 186, 2003.
- [Background] Riggs PD, Hall SK, Mikulich-Gilbertson SK, Lohman M, Kayser A. A randomized controlled trial of pemoline for attention-deficit/hyperactivity disorder in substance-abusing adolescents. J Am Acad Child Adolesc Psychiatry. 2004 Apr;43(4):420-9. doi: 10.1097/00004583-200404000-00008. PMID 15187802
- [Background] Davies RD, Thurstone C, Woyewodzic K. Substance Use Disorders and Neurologic Illness. Curr Treat Options Neurol. 2004 Sep;6(5):421-432. doi: 10.1007/s11940-996-0032-8. PMID 15279762
- [Background] Libby AM, Orton HD, Stover SK, Riggs PD. What came first, major depression or substance use disorder? Clinical characteristics and substance use comparing teens in a treatment cohort. Addict Behav. 2005 Oct;30(9):1649-62. doi: 10.1016/j.addbeh.2005.07.012. Epub 2005 Aug 11. PMID 16098679
- [Background] Libby AM, Riggs PD. Integrated substance use and mental health treatment for adolescents: aligning organizational and financial incentives. J Child Adolesc Psychopharmacol. 2005 Oct;15(5):826-34. doi: 10.1089/cap.2005.15.826. PMID 16262598
- [Background] Drell MJ, Josephson A, Pleak R, Riggs P, Rosenfeld A. Clinical problem solving: the case of John, Part II: excerpts from Sessions 2-7. J Am Acad Child Adolesc Psychiatry. 2006 Oct;45(10):1243-51. doi: 10.1097/01.chi.0000230164.46493.8c. No abstract available. PMID 17003670
- [Background] Thurstone C, Riggs PD, Klein C, Mikulich-Gilbertson SK. A one-session human immunodeficiency virus risk-reduction intervention in adolescents with psychiatric and substance use disorders. J Am Acad Child Adolesc Psychiatry. 2007 Sep;46(9):1179-1186. doi: 10.1097/chi.0b013e31809fe774. PMID 17712241
- [Background] Riggs P. Non-medical use and abuse of commonly prescribed medications. Curr Med Res Opin. 2008 Mar;24(3):869-77. doi: 10.1185/030079908X273435. Epub 2008 Feb 8. PMID 18267053
- [Background] Riggs PD, Mikulich-Gilbertson SK, Davies RD, Lohman M, Klein C, Stover SK. A randomized controlled trial of fluoxetine and cognitive behavioral therapy in adolescents with major depression, behavior problems, and substance use disorders. Arch Pediatr Adolesc Med. 2007 Nov;161(11):1026-34. doi: 10.1001/archpedi.161.11.1026. PMID 17984403
- [Background] Riggs PD, Thompson LL, Tapert SF, Frascella J, Mikulich-Gilbertson S, Dalwani M, Laudenslager M, Lohman M. Advances in neurobiological research related to interventions in adolescents with substance use disorders: research to practice. Drug Alcohol Depend. 2007 Dec 1;91(2-3):306-11. doi: 10.1016/j.drugalcdep.2007.03.003. No abstract available. PMID 18038460